CLINICAL TRIAL: NCT05668156
Title: Defining Fasting: Finding Common Ground Using the Delphi Method
Brief Title: Finding Consensus in Fasting Terminology
Acronym: FT
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: Delphi
Record Dates: First submitted 2022-01-14; First posted 2022-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Consensus Development
Keywords: consensus; fasting; fasting terminology; therapeutic fasting; Delphi; Delphi method; decision-making; intermittent fasting; periodic fasting; prolonged fasting; religious fasting; intermittent dry fasting; caloric restriction; diet; nutrition
MeSH Terms: conditions — Fasting; Intermittent Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Consensus Decision Making — Consensus-based decision-making process, where experts are asked to comment definitions of terms used for fasting interventions

SUMMARY:
A consensus-based decision making process on fasting terminology will be conducted using the Delphi technique. To this aim, experts around the world are invited.

DETAILED DESCRIPTION:
The consensus-based decision making process on fasting terminology will include a maximum of five rounds of questionnaires that experts are invited to complete online using a pseudonym. Prof. Dr. med. Michalsen's department has prepared rough definitions of key terms for the questionnaire to be evaluated by the experts. These terms should serve as a starting point for the discussion. After each questionnaire round the experts' comments are reviewed by the project team and a new questionnaire with the suggested modifications from the previous round will be sent to the experts.

If consensus can't be reached by round three, a live-online-discussion will be held to facilitate the further proceedings.

The results are to be published in a peer-reviewed journal; individual statements will not be shared in the publication.

ELIGIBILITY:
Inclusion Criteria:

* clinicians or scientists with at least 5 peer-reviewed publications on fasting or
* at least one peer-reviewed publication and 5 years of clinical experience with fasting

Exclusion Criteria:

- not more than 2 experts from one institution are allowed to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: clinicians or scientists
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Definitions of fasting regimens | repetition of the survey until consensus is reached, max. 12 months
  Definitions of fasting regimen (qualitative research) with max. five survey rounds and potentially one online discussion panel

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany